CLINICAL TRIAL: NCT04252560
Title: The Impact of Gut Microbiota in Anastomoses Insufficiency After Resection and Direct Anastomosis for Colorectal Cancer.
Status: Completed | Type: Observational
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Tsimogiannis, Principal Investigator, Uppsala University Hospital
Other Study IDs: 2019-04562
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer, Peritoneal Carcinomatosis, Anastomosis Insufficiency
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms | interventions — Colectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal: 30 patients operated for colorectal cancer
  Interventions: Procedure: Colectomy, CRS+HIPEC
- HIPEC: 15 patients operated with CRS+HIPEC for peritoneal carcinomatosis
  Interventions: Procedure: Colectomy, CRS+HIPEC

INTERVENTIONS:
Procedure: Colectomy, CRS+HIPEC — No special interventions are going to be performed. Fecal samples are going to be taken and analysed

SUMMARY:
The role of gut microbiota in anastomosis insufficiency in patients operated for colorectal cancer and for peritoneal carcinomatosis is going to be investigated. This is a pilot study.

ELIGIBILITY:
Inclusion Criteria Colorectal group

* adenocarcinom in colon or rektum
* curative operation planed
* direct anastomose plan
* elective surgery

Inclusion Criteria HIPEC group :

* All patients with appendix, colon or rectal cancer accepted for CRS+HIPEC

Exclusion Criteria:

* Ongoing antibiotics treatment
* antibiotics treatment in the last 6 months
* acute surgery
* palliative surgery
* Ulcerös colitis or Crohns disease
* Prior colectomy
* Small intestine stoma before the operation
* neoadjuvant treatment
* Colon preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the inclusion criteria and have none of the exclusion criteria are going to be asked to participate in the study
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Microbiome | 30 days
  Change in microbiome in case of insufficiency of the anastomosis

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Not allowed by the Ethical Committee